CLINICAL TRIAL: NCT01045759
Title: Intensivist Performed Limited B Mode Compression Ultrasound for Diagnosis of Deep Vein Thrombosis in the Intensive Care Unit
Brief Title: Point of Care Ultrasound (US) Versus Detailed Radiology US for Deep Vein Thrombosis (DVT)
Status: Terminated | Type: Observational
Why Stopped: Investigator left the institution
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: 1143800
Record Dates: First submitted 2010-01-07; First posted 2010-01-11 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: DEEP VEIN THROMBOSIS
Keywords: VENOUS THROMBOSIS; ultrasonography; intensive care unit
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
We propose an observational study to assess the ability of intensivists to evaluate for deep vein thrombosis using 2 point compression ultrasonography.

DETAILED DESCRIPTION:
Deep vein thrombosis is a common problem in the intensive care unit and diagnosis is often delayed due to limited availability of a formal duplex ultrasound. Physician performed 2 point compression ultrasonography has been shown to have reasonable accuracy when performed in the emergency department and outpatient setting, but has not been studied on patients in the intensive care unit. We propose an observational study to assess the ability of intensivists to evaluate for deep vein thrombosis using 2 point compression ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults at least 18 years of age
* Duplex ultrasonography ordered by treating team
* Admission to the Medical, Cardiac, Burn, or Surgical intensive care units

Exclusion Criteria:

* Patients less than 18 years of age
* Patients with a known current DVT
* patients on whom the exam cannot be performed (above the knee amputation, severe cellulitis of groin or popliteal fossa, hip or knee fracture)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients admitted to the intensive care units at University hospital who have a duplex ultrasound of the lower extremities for detection of deep vein thrombosis ordered by the primary team.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2009-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The agreement between physician performed ultrasound and formal duplex ultrasonography for detection of proximal deep vein thrombosis. | 48 hours window from detailed US

SECONDARY OUTCOMES:
Subgroup analysis: location of thrombus (proximal or distal) | 48 hours window from detailed US
Subgroup analysis: number of days in the hospital prior to exam | 48 hours window from detailed US
Subgroup analysis: body mass index (BMI) | 48 hours window from detailed US
Subgroup analysis: weight gain from admission to the time of the exam | 48 hours window from detailed US
Subgroup analysis: training level of examiner | 48 hours window from detailed US
Subgroup analysis: difficulty of exam | 48 hours window from detailed US
Subgroup analysis: specific examiner | 48 hours window from detailed US
Subgroup analysis: presence or absence of calf vein thrombosis | at study conclusion
Subgroup analysis: presence or absence of pulmonary embolism | at study conclusion
Subgroup analysis: DVT location | at study conclusion
Subgroup analysis: calf vein thrombosis | at study conclusion

CONTACTS AND LOCATIONS:
Overall Officials: Casey Stahlheber, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of missouri healthcare, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No